CLINICAL TRIAL: NCT02268526
Title: A Multi-center, Randomized, Double-blind, Placebo Controlled, Study to Evaluate the Efficacy and Safety of CSJ148 Compared to Placebo to Prevent Human Cytomegalovirus (HCMV) Replication in Stem Cell Transplant Patients
Brief Title: Efficacy and Safety Study of CSJ148 in Stem Cell Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCSJ148X2201
Record Dates: First submitted 2014-08-08; First posted 2014-10-20 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: HCMV
Keywords: Safety, efficacy, pharmacokinetics, CSJ148, HCMV, HCMV viral load,; immunogenicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: CSJ148 (Experimental): Cohort 1: CSJ148 IV q 4weeks
  Interventions: Biological: CSJ148
- Cohort 2: CSJ148 (Experimental): Cohort 2: CSJ148 IV q 4weeks
  Interventions: Biological: CSJ148
- Cohort 2: Placebo (Placebo Comparator): Cohort 2: Placebo IV q 4weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSJ148 — CSJ148 IV q 4weeks
  Arms: Cohort 1: CSJ148; Cohort 2: CSJ148
Drug: Placebo — Placebo IV q 4weeks
  Arms: Cohort 2: Placebo

SUMMARY:
This study is designed to test if CSJ148 can prevent HCMV replication after stem cell transplantation.

DETAILED DESCRIPTION:
This study is randomized, double-blinded, and placebo-controlled. 80 Patients will be enrolled and randomized to CSJ148 and placebo in a ratio of 3:1. Patients undergoing stem cell transplantation will be enrolled into the study. The study will consist of a screening period, a baseline visit, approximately 3-month treatment exposure period, an end-of-therapy visit, a follow-up period, and a study completion evaluation approximately 3.5 months after the last dose of study drug is administered.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study had to fulfill all of the following criteria:

1. Written informed consent must be obtained before any assessment was performed.
2. Male and female patients at least 18 years of age.
3. Patients weighed between 45 -120 kg to participate in the study, and had a body mass index (BMI) within the range of 18 - 34 kg/m2
4. Scheduled to undergo allogeneic bone marrow, peripheral blood stem cell, or cord blood transplantation (transplant may be related or unrelated, T-cell depleted or non-T-cell depleted, myeloablative or non-myeloablative/reduced intensity, haploidentical) and began conditioning chemotherapy within 48 hours of planned dosing day.
5. Patient seropositive for HCMV before transplantation; donor could be seropositive or seronegative for HCMV (donor positive/recipient or donor negative/recipient positive). Historical patient HCMV serology data collected within the last 12 months or local assays could be used to qualify the patient for enrollment.
6. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

Patients fulfilling any of the following criteria were not eligible for inclusion in this study:

1. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or until the expected PD (pharmacodynamic) effect has returned to baseline, whichever is longer; or longer if required by local regulations.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
3. Karnofsky performance score <50%.
4. Had HCMV-related organ disease within 6 months prior to enrollment.
5. Detectable HCMV infection (positive pp65 antigenemia or plasma HCMV DNA polymerase chain reaction (PCR) assays prior to enrollment from samples collected within 14 days prior to enrollment. Local assays could be used to qualify the patient for enrollment.
6. Received any of the following within 30 days prior to enrollment: ganciclovir, valganciclovir, foscarnet, cidofovir, acyclovir (>25 mg/kg/day IV), valacyclovir (>3 gm/day oral), famciclovir (>1500 mg/day oral), HCMV immune globulin, immune globulin (>500 mg/kg), or any other medication with anti-HCMV activity.
7. Required mechanical ventilation within 7 days prior to enrollment.
8. Received any vasopressors or other agents for hemodynamic support within 7 days prior to enrollment. These agents included but are not limited to epinephrine, metaraminol, norepinephrine, dopamine, vasopressin, phenylephrine, and dobutamine.
9. Impaired renal function requiring dialysis.
10. Any surgical or medical condition which might increase the risk for thrombotic events if given immunoglobulins. These conditions included cryoglobulinemia, monoclonal gammopathies, and hypertriglyceridemia (fasting level >1000 mg/dL). The investigator should make this determination in consideration of the subject's medical history and laboratory data.
11. Severe liver disease or liver injury as indicated one or more of the following:

    * Alanine aminotransferase (ALT) >5-times the upper limit of normal (ULN).
    * Aspartate aminotransferase (AST) >5-times the upper limit of normal.
    * Gamma-glutamyl transferase (γ-GT) >5-times the upper limit of normal.
    * Serum total bilirubin (TBL) >3-times the upper limit of normal.
12. Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
13. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they were using effective methods of contraception during dosing of study treatment.

    Effective contraception methods included:
    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman was confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that subject.
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository.
    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS). In case of use of oral contraception women would have been stable on the same pill for a minimum of 3 months before taking study treatment. Women were considered post-menopausal and not of child bearing potential if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman had been confirmed by follow up hormone level assessment was she considered not of child bearing potential.
14. History of positive HIV (ELISA and Western blot) test result. Testing was not required. No additional exclusions were applied by the investigator, in order to ensure that the study population was representative of all eligible patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Beech Grove, Indiana
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Houston, Texas
- Novartis Investigative Site, Leuven, Belgium
- Germany (4):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (3):
  - Novartis Investigative Site, New Taipei City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Maertens J, Logan AC, Jang J, Long G, Tang JL, Hwang WYK, Koh LP, Chemaly R, Gerbitz A, Winkler J, Yeh SP, Hiemenz J, Christoph S, Lee DG, Wang PN, Holler E, Mielke S, Akard L, Yeo A, Ramachandra S, Smith K, Pertel P, Segal F. Phase 2 Study of Anti-Human Cytomegalovirus Monoclonal Antibodies for Prophylaxis in Hematopoietic Cell Transplantation. Antimicrob Agents Chemother. 2020 Mar 24;64(4):e02467-19. doi: 10.1128/AAC.02467-19. Print 2020 Mar 24. PMID 32015031
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 1: Six patients were planned for enrollment; 6 patients were enrolled. Cohort 2: Eighty patients were planned and 80 were enrolled.
Period: Overall Study
Arm/Group | Cohort 1: CSJ148 | Cohort 2: CSJ148 | Cohort 2: Placebo
Started | 6 | 59 | 21
PD Analysis Set (Cohort 2) | 0 | 42 | 17
Completed | 5 | 38 | 16
Not Completed | 1 | 21 | 5
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Death | 1 | 11 | 0
Not completed — protocol deviation | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Subject/guardian decision | 0 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: CSJ148 | Cohort 2: CSJ148 | Cohort 2: Placebo | Total
Number analyzed (Participants) | 6 | 59 | 21 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (8.70) | 54.7 (12.33) | 46.0 (14.33) | 52.5 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 23 | 6 | 31
  Male | 4 | 36 | 15 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Require Preemptive HCMV Therapy
Description: Number of participants who require preemptive HCMV therapy. The definition of requiring preemptive anti-HCMV therapy was meeting either one of the following conditions: 1. the plasma HCMV DNA level is >= 1000 copies/mL (with or without HCMV disease) or 2. the plasma HCMV DNA level is < 1000 copies/mL, but HCMV disease was reported
Time Frame: 98 days
Population: Full Analysis Set - included all 86 patients enrolled in the study
Measure: Number; unit: Count of Participants
Groups:
- Total CSJ148 (Cohort 1 & Cohort 2): Cohort 1: CSJ148 IV q 4weeks and Cohort 2: CSJ148 IV q 4weeks
Arm/Group | Total CSJ148 (Cohort 1 & Cohort 2) | Cohort 2: CSJ148 | Cohort 2: Placebo
Number analyzed (Participants) | 65 | 59 | 21
Count of Participants | 24 | 23 | 9
Statistical Analysis 1: Comparison: Total CSJ148 (Cohort 1 & Cohort 2) vs Cohort 2: Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 0.891, 90% CI 2-sided [0.606 to 1.305]
Statistical Analysis 2: Comparison: Cohort 2: CSJ148 vs Cohort 2: Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 0.941, 90% CI 2-sided [0.639 to 1.377]

2. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Number of participants with adverse events as a measure of safety and tolerability. Patients treated with CSJ148 in Cohorts 1 and 2 were pooled to simplify the safety analyses.
Time Frame: 98 days
Population: Safety Analysis Set- Eighty-six patients were enrolled in the study and all were included in the safety analysis set
Measure: Number; unit: Count of Participants
Groups:
- Total CSJ148 (Cohort 1 & Cohort 2): Cohort 1: CSJ148 IV q 4weeks & Cohort 2: CSJ148 IV q 4 weeks
Arm/Group | Total CSJ148 (Cohort 1 & Cohort 2) | Cohort 2: Placebo
Number analyzed (Participants) | 65 | 21
Count of Participants
  At least one treatment-emergent AE | 65 | 21
  At least one drug-related AE | 0 | 2
  At least one SAE | 46 | 15
  At least one drug-related SAE | 0 | 1
  Deaths | 12 | 0
  At least 1 treatment-emergent AE grade 3 or higher | 58 | 17
  Total deaths:those reported after study completion | 19 | 3
  Discontinued study treatment due to any AE | 1 | 1

3. Secondary Outcome: Time to Start of Preemptive HCMV Therapy Cohort 2
Description: The time to start preemptive therapy is defined as the number of days between initial dose of study drug and the earlier of (1) the start of preemptive therapy, and (2) the development of HCMV disease or death due to HCMV disease, or (3) censored at the EoT visit if no therapy required for Cohort 2
Time Frame: 98 days
Population: PD analysis set (Cohort 2) -included 59 patients, 27 patients (31%) were excluded.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 2: CSJ148 | Cohort 2: Placebo
Number analyzed (Participants) | 42 | 17
days | 62.03 (12.145) | 49.54 (13.470)

4. Secondary Outcome: Number of Times That Preemptive HCMV Therapy is Required -Cohort 2
Description: Among those who required preemptive therapy, the number of times preemptive therapy was required. (Cohort 2)
Time Frame: 98 days
Population: PD analysis set (Cohort 2) -included 59 patients, 27 patients (31%) were excluded.
Measure: Least Squares Mean (90% Confidence Interval); unit: number of times
Arm/Group | Cohort 2: CSJ148 | Cohort 2: Placebo
Number analyzed (Participants) | 42 | 17
number of times | 2.070 [1.369 to 3.130] | 2.540 [1.342 to 4.806]

5. Secondary Outcome: Proportion of Participants Developing HCMV Disease
Description: Proportion of participants developing HCMV disease
Time Frame: 98 days
Population: PD analysis set (Cohort 2) -included 59 patients, 27 patients (31%) were excluded.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 2: CSJ148 | Cohort 2: Placebo
Number analyzed (Participants) | 42 | 17
proportion of participants | 0.119 [0.048 to 0.234] | 0 [0 to 0.162]

6. Secondary Outcome: Area Under the Serum Concentration-time Curve During the Dosing Interval (AUCtau) for CSJ148 Only
Description: PK parameters were calculated from plasma concentration-time data using non-compartmental methods. The AUCtau was calculated using a linear trapezoidal method
Time Frame: Day 1, Day 29, Day 57, Day 85 at predose (0hr) and 3,6,24 hrs post dose
Population: Pharmacokinetics (PK) analysis set (CSJ148 only)- The PK analysis set included the 65 patients who received a dose of CSJ148
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Total CSJ148 (Cohort 1 & Cohort 2)
Number analyzed (Participants) | 65
day*ug/mL
  Day 1 | 7310 (2310)
  Day 29 | 9890 (3470)
  Day 57 | 11400 (4020)
  Day 85 | 12900 (4380)

7. Secondary Outcome: Maximum Serum Concentration During the Dosing Interval (Cmax) for CSJ148 Only
Description: Cmax is the observed maximum plasma (or serum or blood) concentration following drug administration [ug / mL] for CSJ148 only
Time Frame: Day 1, Day 29, Day 57, Day 85 at predose (0hr) and 3,6,24 hrs post dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Total CSJ148 (Cohort 1 & Cohort 2)
Number analyzed (Participants) | 65
ug/mL
  Day 1 | 1040 (356)
  Day 29 | 1100 (282)
  Day 57 | 1180 (316)
  Day 85 | 1230 (458)

8. Secondary Outcome: Trough Serum Concentration (Ctrough) for CSJ148 Only
Description: Ctrough is The observed plasma (or serum or blood) concentration at the end of a drug administration dosing interval [ug / mL]
Time Frame: Day 1, Day 29, Day 57, Day 85 at predose (0hr) and 3,6,24 hrs post dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Total CSJ148 (Cohort 1 & Cohort 2)
Number analyzed (Participants) | 65
ug/mL
  Day 1 | 104 (59.7)
  Day 29 | 167 (85.5)
  Day 57 | 214 (152)
  Day 85 | 223 (104)

9. Secondary Outcome: Accumulation Ratio(Racc) for CSJ148 Only at Day 85
Description: Accumulation ratio(Racc) is Racc: Accumulation ratio, calculated by AUCtau (Day 85) divided by AUCtau (for the 1st dose at Day 1).
Time Frame: Day 1 and Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Total CSJ148 (Cohort 1 & Cohort 2)
Number analyzed (Participants) | 65
Ratio | 1.83 (0.531)

10. Secondary Outcome: Lambda_z for CSJ148 Only at Day 85
Description: Lambda_z is the terminal elimination rate constant [1/day] at Day 85
Time Frame: Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1/day
Arm/Group | Total CSJ148 (Cohort 1 & Cohort 2)
Number analyzed (Participants) | 65
1/day | 0.0409 (0.0175)

11. Secondary Outcome: Half-life (T1/2) for CSJ148 Only at Day 85
Description: T1/2 is the terminal elimination half-life [time]
Time Frame: Day 85
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: day
Arm/Group | Total CSJ148 (Cohort 1 & Cohort 2)
Number analyzed (Participants) | 65
day | 19.7 (7.18)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit 183 days.
Description: Additional 2 deaths in placebo occurred during follow-up (Day 100 to 183) after early treatment and study discontinuation. One additional placebo death occurred after end of study (Day 183) and 7 additional CSJ148 deaths occurred post end of study (Day 183).
  Patients treated with CSJ148 in Cohorts 1 and 2 were pooled to simplify the safety analyses because the dosage of CSJ148 was the same for each cohort. Cohort 1 was just a PK cohort with only 6 patients.
Groups:
- Placebo: Cohort 2: Placebo IV q 4weeks
- Total CSJ148: Cohort 1: CSJ148 IV q 4weeks & Cohort 2: CSJ148 IV q 4weeks
Arm/Group | Placebo | Total CSJ148
Serious Adverse Events (participants affected / at risk) | 15/21 | 46/65
Other Adverse Events (participants affected / at risk) | 21/21 | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Total CSJ148 (N=65)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 8
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Splenic lesion (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Intracardiac mass (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis erosive (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal lesion (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 3
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Acute graft versus host disease (Immune system disorders) | 2 | 9
Acute graft versus host disease in liver (Immune system disorders) | 0 | 1
Acute graft versus host disease in skin (Immune system disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Chronic graft versus host disease in liver (Immune system disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 2
Cytomegalovirus gastritis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 2
Cytomegalovirus viraemia (Infections and infestations) | 2 | 2
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 0 | 1
Epididymitis tuberculous (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
JC virus infection (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 4
Septic shock (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Stenotrophomonas infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Engraft failure (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Cytomegalovirus test positive (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Chronic myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 4
Renal disorder (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Total CSJ148 (N=65)
Anaemia (Blood and lymphatic system disorders) | 4 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 25
Neutropenia (Blood and lymphatic system disorders) | 5 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 9
Tachycardia (Cardiac disorders) | 2 | 8
Dry eye (Eye disorders) | 5 | 14
Abdominal discomfort (Gastrointestinal disorders) | 1 | 6
Abdominal distension (Gastrointestinal disorders) | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 5 | 16
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 8 | 19
Diarrhoea (Gastrointestinal disorders) | 12 | 43
Dry mouth (Gastrointestinal disorders) | 3 | 11
Dyspepsia (Gastrointestinal disorders) | 3 | 7
Epigastric discomfort (Gastrointestinal disorders) | 2 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 6
Haemorrhoids (Gastrointestinal disorders) | 2 | 13
Lip dry (Gastrointestinal disorders) | 2 | 1
Melaena (Gastrointestinal disorders) | 0 | 4
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 14 | 45
Oesophagitis (Gastrointestinal disorders) | 1 | 9
Stomatitis (Gastrointestinal disorders) | 15 | 36
Tongue ulceration (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 14 | 38
Asthenia (General disorders) | 2 | 7
Catheter site erythema (General disorders) | 2 | 4
Catheter site pain (General disorders) | 1 | 6
Chest discomfort (General disorders) | 1 | 5
Chills (General disorders) | 4 | 15
Fatigue (General disorders) | 7 | 18
Generalised oedema (General disorders) | 0 | 7
Non-cardiac chest pain (General disorders) | 1 | 8
Oedema peripheral (General disorders) | 2 | 12
Pain (General disorders) | 0 | 6
Pyrexia (General disorders) | 10 | 38
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 4
Acute graft versus host disease (Immune system disorders) | 3 | 10
Acute graft versus host disease in intestine (Immune system disorders) | 0 | 4
Acute graft versus host disease in skin (Immune system disorders) | 3 | 14
Chronic graft versus host disease (Immune system disorders) | 4 | 6
Chronic graft versus host disease in skin (Immune system disorders) | 1 | 5
Candida infection (Infections and infestations) | 0 | 5
Clostridium difficile infection (Infections and infestations) | 0 | 5
Device related infection (Infections and infestations) | 2 | 3
Folliculitis (Infections and infestations) | 2 | 7
Herpes zoster (Infections and infestations) | 2 | 4
Human herpesvirus 6 infection (Infections and infestations) | 1 | 4
Oral candidiasis (Infections and infestations) | 3 | 5
Oral herpes (Infections and infestations) | 1 | 4
Papilloma viral infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 4
Rhinovirus infection (Infections and infestations) | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 8
Urinary tract infection (Infections and infestations) | 1 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 6
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 4
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 5
Alanine aminotransferase increased (Investigations) | 2 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 4
Blood bilirubin increased (Investigations) | 1 | 7
Blood creatinine increased (Investigations) | 3 | 8
Decreased appetite (Metabolism and nutrition disorders) | 7 | 27
Fluid overload (Metabolism and nutrition disorders) | 1 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 20
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 17
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Dizziness (Nervous system disorders) | 3 | 16
Headache (Nervous system disorders) | 6 | 24
Neuropathy peripheral (Nervous system disorders) | 1 | 6
Syncope (Nervous system disorders) | 0 | 4
Tremor (Nervous system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 0 | 5
Confusional state (Psychiatric disorders) | 0 | 7
Hallucination (Psychiatric disorders) | 0 | 5
Insomnia (Psychiatric disorders) | 6 | 15
Sleep disorder (Psychiatric disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 5
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 2 | 5
Haematuria (Renal and urinary disorders) | 1 | 10
Pollakiuria (Renal and urinary disorders) | 2 | 8
Scrotal pain (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 12
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 6
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 18
Rash (Skin and subcutaneous tissue disorders) | 7 | 24
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 6
Hypertension (Vascular disorders) | 5 | 23
Hypotension (Vascular disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single- site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.